CLINICAL TRIAL: NCT05371652
Title: A Multicenter, Open Label, Long-term Safety Study of BHV3000 for the Acute Treatment of Migraine in Chinese Subjects
Brief Title: A Study to Learn About the Long-term Safety of Rimegepant for the Acute Treatment of Migraine in Chinese Participants
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BHV3000-318; C4951018 (Other: Alias Study Number)
Record Dates: First submitted 2022-03-23; First posted 2022-05-12 (Actual); Results first posted 2025-02-20 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-01

CONDITIONS: Acute Migraine
Keywords: Migraine
MeSH Terms: conditions — Migraine Disorders | interventions — rimegepant sulfate

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Rimegepant 75mg Orally Disintegrating Tablets (ODT) (Experimental): One rimegepant (BHV3000) 75mg orally disintegrating tablet (up to 1 tablet per day)
  Interventions: Drug: Rimegepant 75mg Orally Disintegrating Tablets (ODT)

INTERVENTIONS:
Drug: Rimegepant 75mg Orally Disintegrating Tablets (ODT) — One rimegepant (BHV3000) 75mg orally disintegrating tablet (up to 1 tablet per day) at the time of their migraine attack

SUMMARY:
This trial is to evaluate the long-term safety and tolerability of Rimegepant 75mg ODT in Chinese subjects with migraine

ELIGIBILITY:
Inclusion Criteria:

At least a one-year history of migraines (with or without aura), consistent with a diagnosis according to the International Classification of Headache Disorders, 3rd edition beta version, including the following:

* Age of onset of migraines prior to 50 years of age
* Migraine attacks, on average, lasting 4 - 72 hours if untreated
* 6-18 migraine attacks of moderate or severe intensity per month within the last 3 months prior to the Screening Visit
* 6 or more migraine days requiring treatment during Observation Phase
* Ability to distinguish migraine attacks from tension/cluster headaches
* Subjects on prophylactic migraine medication are permitted to remain on therapy if the dose has been stable dose for at least 2 months prior to the Baseline Visit, and the dose is not expected to change during the course of the study. subjects who previously discontinued prophylactic migraine medication must have done so at least 5 half-lives of the prophylactic medication prior to the Screening Visit
* Subjects with contraindications for use of triptans may be included provided they meet all other study entry criteria

Age and Reproductive Status:

* Male or female subjects ≥ 18 years
* Women of childbearing potential (WOCBP) must voluntarily use 1 acceptable methods of contraception to avoid pregnancy and to minimize the risk of pregnancy from signing of informed consent through 28 days after study drug administration. WOCBP is defined in Section 12.3. No contraception methods are required for male subjects in this study.

Exclusion Criteria:

Target Disease Exclusion:

* Subjects has a history of basilar migraine with brain stem aura or hemiplegic migraine

Medical History and Comorbidities:

* History of HIV disease
* Current evidence of poorly controlled, unstable, or recently diagnosed cardiovascular or cerebrovascular disease such as ischemic heart disease, coronary vasospasm, and cerebral ischemia. Myocardial infarction (MI), acute coronary syndrome (ACS), percutaneous coronary intervention (PCI), cardiac surgery, stroke, or transient ischemic attack (TIA) during 6 months prior to screening
* Poorly controlled hypertension (high blood pressure) or poorly controlled diabetes (but subjects with stable hypertension and/or diabetes for at least 3 months prior to screening may be included in the study). Blood pressure greater than 150 mmHg systolic or 100 mmHg diastolic after 10 minutes of rest is exclusionary
* Subjects with a current diagnosis of major depression or a major depressive episode within the last 12 months, other pain syndromes, psychiatric disorders, dementia, or significant neurological disorders (other than migraine) that, in the opinion of the investigator, might interfere with study assessments
* History of gastric or small intestinal surgery (including gastric bypass, gastric banding, gastric sleeve, gastric water ball, etc.) or diseases resulting in malabsorption
* Subject has a history or diagnosis of Gilibert's Syndrome or any other active hepatic or biliary disorder
* History or presence of significant and/or unstable medical conditions (e.g., history of congenital heart disease or cardiac arrhythmia, known suspected infection, hepatitis B or C or neoplasm) that, in the opinion of the investigator, would expose the subjects to undue risk of a significant adverse events (AE) or interfere with the assessment of safety or effectiveness during the trial
* History or evidence of alcohol or drug abuse within the past 12 months, or treatment for alcohol or drug abuse, or meeting Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-V) criteria for any significant substance abuse disorder within the past 12 months prior to the Screening Visit
* Subjects should be excluded if they have a positive drug screen for drugs of abuse and are considered medically significant by the investigator, would compromise subject safety, or interfere with the interpretation of study results. In addition:
* Subjects with detectable levels of cocaine, amphetamines, and phencyclidine in drug abuse screening need to be excluded.

Subjects who are positive for amphetamines on the urine drug screen may have their urine samples evaluated for further analysis at the investigator's discretion to rule out a false positive result

* Subjects with detectable levels of marijuana during substance abuse screening may not be excluded if they do not meet DSMV criteria for substance abuse or dependence in the subject's opinion as documented by the investigator, and a positive result does not signal a clinical condition that would impact the subject safety or interpretation of the study results
* Diagnosis of hematologic or solid malignancy within 5 years prior to screening. Subjects with a history of localized basal cell or squamous cell skin cancer may be included in the study if they are cancer-free prior to the screening visit for this study
* Subjects with a current diagnosis of schizophrenia, major depression requiring treatment with atypical antipsychotics, bipolar disorder or borderline personality disorder
* Body mass index (BMI) ≥ 35 kg/ m2
* Subjects with a history of gallstones or cholecystectomy
* Use of St. John's Wort, products containing St. John's Wort, Coltsfoot root, or extracts within 14 days prior to the baseline visit
* Use of narcotic drugs such as opioids (e.g., morphine, codeine, oxycodone, and hydrocodone) within 2 days prior to the baseline visit.

Allergy and Adverse Reactions:

*. History of drug or other allergy that, in the opinion of the investigator, would make the subject unsuitable for participation in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 241 (Actual)
Dates: Start 2022-05-19 (Actual); Primary Completion 2024-02-06 (Actual); Study Completion 2024-02-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (25):
- China (25):
  - The Second Hospital of Anhui Medical University, Hefei, Anhui
  - Beijing Friendship Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Chinese PLA General Hospital, Beijing, Beijing Municipality
  - The First Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality
  - The First Affiliated hospital of Xiamen University, Xiamen, Fujian
  - Hainan General Hospital, Haikou, Hainan
  - Hebei General Hospital, Shijiazhuang, Hebei
  - Renmin Hospital Of Wuhan University, Wuhan, Hubei
  - Wuhan Third Hospital, Wuhan, Hubei
  - Changsha Central Hospital, Changsha, Hunan
  - Xiangya Hospital Central South University, Changsha, Hunan
  - The Third Xiangya Hospital of Central South University, Changsha, Hunan
  - The Second Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu
  - The Second Hospital of Jilin University, Changchun, Jilin
  - General Hospital of Northern Theater Command, Shenyang, Liaoning
  - Shaanxi Provincial People' Hospital, Xi'an, Shaanxi
  - The First Affiliated Hospital of Xi'an Medical University, Xi'an, Shaanxi
  - Yan'an University Xianyang Hospital Co., Ltd, Xianyang, Shaanxi
  - LiaoCheng People's Hospital, Liaocheng, Shandong
  - Tongji Hospital of Tongji University, Shanghai, Shanghai Municipality
  - West China Hospital of Sichuan University, Chengdu, Sichuan
  - The Second Affiliated Hospital of Xinjiang Medical University, Ürümqi, Xinjiang
  - The Second Affiliated hospital of Kunming Medical University, Kunming, Yunnan
  - Peking University People's Hospital, Beijing
  - Guangzhou First People's Hospital, Guangzhou

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- [Derived] Zhang M, Guo A, Wu J, Wang H, Zhang Y, Dong H, Liu J, Zhang B, Guo H, Yu T, Lu Z, Ma L, Fountaine RJ, Pixton GC, Zhong Q, Han X, Yu S. Rimegepant for the acute treatment of migraine: A phase 3, multicenter, open-label, long-term safety and effectiveness study in adults from China. Cephalalgia. 2025 Oct;45(10):3331024251371686. doi: 10.1177/03331024251371686. Epub 2025 Oct 9. PMID 41066271
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=BHV3000-318

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 241 participants were enrolled in the study. 240 participants received study treatment.
Groups:
- Rimegepant 75 Milligrams (mg) Orally Disintegrating Tablets (ODT): Chinese participants with migraine received 75 mg of rimegepant ODT (Pro re nata [PRN] use, up to 1 tablet per day) for 52 weeks.
Period: Overall Study
Arm/Group | Rimegepant 75 Milligrams (mg) Orally Disintegrating Tablets (ODT)
Started | 241
Treated | 240
Completed | 208
Not Completed | 33
Not completed — Non-Compliance with Study Schedule | 9
Not completed — Withdrawal by Subject | 12
Not completed — Adverse Event | 1
Not completed — Other | 11

BASELINE CHARACTERISTICS:
Population: Full Analysis set included all participants who were enrolled and received at least one dose of the investigational product.
Groups:
- Rimegepant 75mg ODT: Chinese participants with migraine received 75 mg of rimegepant ODT (PRN use, up to 1 tablet per day) for 52 weeks.
Arm/Group | Rimegepant 75mg ODT
Number analyzed (Participants) | 240
Age, Continuous [Mean (Standard Deviation); unit: Years] | 39.1 (10.97)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 192
  Male | 48
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 240
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Han | 231
  Unknown or not reported | 9

OUTCOME MEASURES:

1. Primary Outcome: Treatment Safety Period: Number of Participants With Treatment Emergent Adverse Events (TEAEs)
Description: An adverse event was any untoward medical occurrence in a clinical trial participant administered an investigational product that may present with symptoms/signs, disease, or laboratory abnormalities and which did not necessarily have a causal relationship with the investigational product. TEAEs were events that started after the first dose of trial drug and did not occur or worsen relative to the first dose.
Time Frame: From Day 1 of study treatment up to Week 52 of the treatment safety period
Population: Safety analysis set (SS) included all participants who received at least one dose of investigational product.
Measure: Count of Participants; unit: Participants
Groups:
- Rimegepant 75 mg ODT: Chinese participants with migraine received 75 mg of rimegepant ODT (PRN use, up to 1 tablet per day) for 52 weeks.
Arm/Group | Rimegepant 75 mg ODT
Number analyzed (Participants) | 240
Participants | 203

2. Primary Outcome: Follow-up Safety Period: Number of Participants With TEAEs
Description: as for outcome 1
Time Frame: From Week 52 to Week 54 of the follow-up safety period
Population: Follow-up safety analysis set (FUSS) included all participants in the SS with last contact date in the follow-up safety analysis period.
Measure: Count of Participants; unit: Participants
Arm/Group | Rimegepant 75 mg ODT
Number analyzed (Participants) | 228
Participants | 24

3. Primary Outcome: Treatment Safety Period: Number of Participants With Serious Adverse Events (SAEs)
Description: An adverse event was any untoward medical occurrence in a clinical trial participant administered an investigational product that may present with symptoms/signs, disease, or laboratory abnormalities and which did not necessarily have a causal relationship with the investigational product. SAE referred to any untoward medical occurrence that met any of the following criteria at any dose for a participant that received the investigational product: death, life-threatening, permanent or severe disability or incapacity, hospitalization or prolongation of hospitalization required or congenital anomaly or birth defect.
Time Frame: From Day 1 of study treatment up to Week 52 of the treatment safety period
Population: Safety analysis set included all participants who received at least one dose of investigational product.
Measure: Count of Participants; unit: Participants
Arm/Group | Rimegepant 75 mg ODT
Number analyzed (Participants) | 240
Participants | 7

4. Primary Outcome: Follow-up Safety Period: Number of Participants With SAEs
Description: as for outcome 3
Time Frame: From Week 52 to Week 54 of the follow-up safety period
Population: FUSS included all participants in the SS with last contact date in the follow-up safety analysis period.
Measure: Count of Participants; unit: Participants
Arm/Group | Rimegepant 75 mg ODT
Number analyzed (Participants) | 228
Participants | 0

5. Primary Outcome: Treatment Safety Period: Number of Participants With AEs Leading to Study Drug Discontinuation
Description: An AE was any untoward medical occurrence in a clinical trial participant administered an investigational product that may present with symptoms/signs, disease, or laboratory abnormalities and which did not necessarily had a causal relationship with the investigational product. AEs that led to study drug discontinuation were reported in this outcome measure.
Time Frame: From Day 1 of study treatment up to Week 52 of the treatment safety period
Population: Safety analysis set included all participants who received at least one dose of investigational product.
Measure: Count of Participants; unit: Participants
Arm/Group | Rimegepant 75 mg ODT
Number analyzed (Participants) | 240
Participants | 1

6. Primary Outcome: Follow-up Safety Period: Number of Participants With AEs Leading to Study Drug Discontinuation
Description: as for outcome 5
Time Frame: From Week 52 to Week 54 of the follow-up safety period
Population: FUSS included all participants in the SS with last contact date in the follow-up safety analysis period.
Measure: Count of Participants; unit: Participants
Arm/Group | Rimegepant 75 mg ODT
Number analyzed (Participants) | 228
Participants | 0

7. Primary Outcome: Treatment Safety Period: Number of Participants With Electrocardiogram (ECG) Abnormalities
Description: ECG abnormalities criteria included: QT Interval Corrected Using Fridericia's Formula (QTcF) millisecond (msec): less than or equal to (<=)450, 450 - <=480, 480- <=500, greater than (>)500.
Time Frame: From Day 1 of study treatment up to Week 52 of the treatment safety period
Population: Safety analysis set included all participants who received at least one dose of investigational product.
Measure: Count of Participants; unit: Participants
Arm/Group | Rimegepant 75 mg ODT
Number analyzed (Participants) | 240
Participants
  <=450 | 225
  450 - <= 480 | 6
  480 - <= 500 | 0
  > 500 | 0

8. Primary Outcome: Follow-up Safety Period: Number of Participants With ECG Abnormalities
Description: ECG abnormalities criteria included: QTcF msec: <=450, 450 - <=480, 480- <=500, >500.
Time Frame: From Week 52 to Week 54 of the follow-up safety period
Population: FUSS included all participants in the SS with last contact date in the follow-up safety analysis period.
Measure: Count of Participants; unit: Participants
Arm/Group | Rimegepant 75 mg ODT
Number analyzed (Participants) | 228
Participants
  <=450 | 209
  450 - <= 480 | 2
  480 - <= 500 | 0
  >500 | 2

9. Primary Outcome: Treatment Safety Period: Number of Participants With Vital Signs Abnormalities
Description: Vital signs abnormalities included blood pressure (BP) millimeters of mercury (mmHg): systolic BP <90 and >140; diastolic BP <50 and >90 and pulse rate (beats per minute) :<40 and >120.
Time Frame: From Day 1 of study treatment up to Week 52 of the treatment safety period
Population: Safety analysis set included all participants who received at least one dose of investigational product. Here, "Number of Participants Analyzed" signifies participants evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Rimegepant 75 mg ODT
Number analyzed (Participants) | 238
Participants
  Systolic BP <90 | 12
  Systolic BP >140 | 9
  Diastolic BP <50 | 1
  Diastolic BP >90 | 17
  Pulse rate <40 | 0
  Pulse rate >120 | 0

10. Primary Outcome: Follow-up Safety Period: Number of Participants With Vital Signs Abnormalities.
Description: Vital signs abnormalities included BP mmHg: systolic BP <90 and >140; diastolic BP <50 and >90 and pulse rate (beats per minute) :<40 and >120.
Time Frame: From Week 52 to Week 54 of the follow-up safety period
Population: FUSS included all participants in the SS with last contact date in the follow-up safety analysis period. Here, "Number of Participants Analyzed" signifies participants evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Rimegepant 75 mg ODT
Number analyzed (Participants) | 213
Participants
  Systolic BP <90 | 1
  Systolic BP >140 | 1
  Diastolic BP <50 | 0
  Diastolic BP >90 | 5
  Pulse rate <40 | 0
  Pulse rate >120 | 0

11. Primary Outcome: Treatment Safety Period: Number of Participants With Hematology Test Abnormalities
Description: Hematology parameters included: hemoglobin increased, anemia, leukocytosis, white blood cell decreased, platelet count decreased, neutrophil count decreased, lymphocyte count increased, lymphocyte count decreased. As per National Cancer Institute of Common Terminology Criteria for Adverse Events (NCI CTCAE) version(v)5.0-Grade(G) 1: mild; asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated, Grade 2: moderate; minimal, local or non-invasive intervention indicated; limiting age appropriate instrumental activities of daily living (ADL), Grade 3: severe or medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; limiting self-care ADL. Grade 4: life-threatening consequences; urgent intervention indicated. Grade 5: death related to AE. Grade 3 and 4 abnormalities were reported in this outcome measure.
Time Frame: From Day 1 of study treatment up to Week 52 of the treatment safety period
Population: Safety analysis set included all participants who received at least one dose of investigational product.
Measure: Count of Participants; unit: Participants
Arm/Group | Rimegepant 75 mg ODT
Number analyzed (Participants) | 240
Participants
  Hemoglobin increased | 0
  Anemia | 1
  Leukocytosis | 0
  White blood cell decreased | 1
  Platelet count decreased | 0
  Neutrophil count decreased | 1
  Lymphocyte count increased | 0
  Lymphocyte count decreased | 1

12. Primary Outcome: Follow-up Safety Period: Number of Participants With Hematology Test Abnormalities
Description: Hematology parameters included: hemoglobin increased, anemia, leukocytosis, white blood cell decreased, platelet count decreased, neutrophil count decreased, lymphocyte count increased, lymphocyte count decreased. As per NCI CTCAE v5.0-Grade 1: mild; asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated, Grade 2: moderate; minimal, local or non-invasive intervention indicated; limiting age-appropriate instrumental ADL, Grade 3: severe or medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; limiting self-care ADL. Grade 4: life-threatening consequences; urgent intervention indicated. Grade 5: death related to AE. Grade 3 and 4 abnormalities were reported in this outcome measure.
Time Frame: From Week 52 to Week 54 of the follow-up safety period
Population: FUSS included all participants in the SS with last contact date in the follow-up safety analysis period.
Measure: Count of Participants; unit: Participants
Arm/Group | Rimegepant 75 mg ODT
Number analyzed (Participants) | 228
Participants
  Hemoglobin increased | 0
  Anemia | 0
  Leukocytosis | 0
  White blood cell decreased | 0
  Platelet count decreased | 0
  Neutrophil count decreased | 1
  Lymphocyte count increased | 0
  Lymphocyte count decreased | 0

13. Primary Outcome: Treatment Safety Period: Number of Participants With Chemistry Test Abnormalities
Description: Chemistry Test Abnormalities included: hypernatremia, hyponatremia, hyperkalemia, hypokalemia, hypoglycemia, creatinine increased, blood lactate dehydrogenase increased, hypoalbuminemia, creatine phosphokinase (CPK) increased, aspartate aminotransferase increased, alanine aminotransferase increased, blood bilirubin increased, alkaline phosphatase increased, chronic kidney disease, cholesterol high, hypertriglyceridemia. As per NCI CTCAE v5.0-G1: mild; asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated, G2: moderate; minimal, local or non-invasive intervention indicated; limiting age-appropriate instrumental ADL, G3: severe or medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; limiting self-care ADL. G4: life-threatening consequences; urgent intervention indicated. G5: death related to AE. G3 and 4 abnormalities were reported in this outcome measure.
Time Frame: From Day 1 of study treatment up to Week 52 of the treatment safety period
Population: Safety analysis set included all participants who received at least one dose of investigational product.
Measure: Count of Participants; unit: Participants
Arm/Group | Rimegepant 75 mg ODT
Number analyzed (Participants) | 240
Participants
  Hypernatremia | 0
  Hyponatremia | 0
  Hyperkalemia | 0
  Hypokalemia | 1
  Hypoglycemia | 0
  Creatinine increased | 0
  Blood lactate dehydrogenase increased | 0
  Hypoalbuminemia | 0
  CPK increased | 4
  Aspartate aminotransferase increased | 1
  Alanine aminotransferase increased | 0
  Blood bilirubin increased | 0
  Alkaline phosphatase increased | 0
  Chronic kidney disease | 0
  Cholesterol high | 0
  Hypertriglyceridemia | 2

14. Primary Outcome: Follow-up Safety Period: Number of Participants With Chemistry Test Abnormalities
Description: Chemistry Test Abnormalities included: hypernatremia, hyponatremia, hyperkalemia, hypokalemia, hypoglycemia, creatinine increased, blood lactate dehydrogenase increased, hypoalbuminemia, CPK increased, aspartate aminotransferase increased, alanine aminotransferase increased, blood bilirubin increased, alkaline phosphatase increased, chronic kidney disease, cholesterol high, hypertriglyceridemia. As per NCI CTCAE v5.0-G1: mild; asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated, G2: moderate; minimal, local or non-invasive intervention indicated; limiting age-appropriate instrumental ADL, G3: severe or medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; limiting self-care ADL. G4: life-threatening consequences; urgent intervention indicated. Grade 5: death related to AE. G3 and 4 abnormalities were reported in this outcome measure.
Time Frame: From Week 52 to Week 54 of the follow-up safety period
Population: FUSS included all participants in the SS with last contact date in the follow-up safety analysis period.
Measure: Count of Participants; unit: Participants
Arm/Group | Rimegepant 75 mg ODT
Number analyzed (Participants) | 228
Participants
  Hypernatremia | 0
  Hyponatremia | 0
  Hyperkalemia | 0
  Hypokalemia | 1
  Hypoglycemia | 0
  Creatinine increased | 0
  Blood lactate dehydrogenase increased | 0
  Hypoalbuminemia | 0
  CPK increased | 0
  Aspartate aminotransferase increased | 0
  Alanine aminotransferase increased | 0
  Blood bilirubin increased | 0
  Alkaline phosphatase increased | 0
  Chronic kidney disease | 0
  Cholesterol high | 0
  Hypertriglyceridemia | 0

15. Secondary Outcome: Change From Observation Period in the Number of Migraine Days by Pain Intensity at Every 4 Week Interval and Overall Period
Description: The number of migraine days and severity of migraine attacks was analyzed for every 4-week interval and overall period during long-term treatment with rimegepant in participants was compared to the observation period. Pain intensity of migraine was graded into mild, moderate, or severe and severity was judged by investigator.
Time Frame: Baseline (observation period); Week 1 to 4, 5 to 8, 9 to 12, 13 to 16, 17 to 20, 21 to 24, 25 to 28, 29 to 32, 33 to 36, 37 to 40, 41 to 44, 45 to 48, 49 to 52 and Overall (Week 1 to 52)
Population: Efficacy analysis set (EAS) included all participants in the FAS with>= 14 electronic (e)Diary days (not necessarily consecutive) in both the observational period analysis period and>= 1 month (4-week interval) of the long-term treatment analysis period. "Number Analyzed" signifies number of participants evaluable for the specified rows.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Rimegepant 75 mg ODT
Number analyzed (Participants) | 240
Days
  Week 1 to Week 4 | -1.7 (3.8)
  Week 5 to Week 8: number analyzed (Participants) | 236
  Week 5 to Week 8 | -2.4 (4.5)
  Week 9 to Week 12: number analyzed (Participants) | 233
  Week 9 to Week 12 | -3.4 (4.2)
  Week 13 to Week 16: number analyzed (Participants) | 229
  Week 13 to Week 16 | -3.7 (4.6)
  Week 17 to Week 20: number analyzed (Participants) | 228
  Week 17 to Week 20 | -4.4 (4.6)
  Week 21 to Week 24: number analyzed (Participants) | 224
  Week 21 to Week 24 | -4.8 (4.6)
  Week 25 to Week 28: number analyzed (Participants) | 221
  Week 25 to Week 28 | -5.2 (4.6)
  Week 29 to Week 32: number analyzed (Participants) | 219
  Week 29 to Week 32 | -4.8 (4.7)
  Week 33 to Week 36: number analyzed (Participants) | 218
  Week 33 to Week 36 | -5.2 (4.5)
  Week 37 to Week 40: number analyzed (Participants) | 215
  Week 37 to Week 40 | -5.5 (5.1)
  Week 41 to Week 44: number analyzed (Participants) | 213
  Week 41 to Week 44 | -5.7 (4.7)
  Week 45 to Week 48: number analyzed (Participants) | 211
  Week 45 to Week 48 | -5.6 (4.7)
  Week 49 to Week 52: number analyzed (Participants) | 207
  Week 49 to Week 52 | -5.6 (5.5)
  Overall | -2.8 (4.1)

ADVERSE EVENTS:
Time Frame: From Day 1 of study treatment up to Week 54
Description: Same event may appear as both non-SAE and SAE but what is presented are distinct events. An event may be categorized as serious in one participant and non-serious in another participant or one participant may have experienced both serious and non-serious event. Safety analysis set included all participants who received at least one dose of investigational product. The SS used for safety analyses during treatment safety period.
Arm/Group | Rimegepant 75 mg ODT
All-Cause Mortality (participants affected / at risk) | 1/240
Serious Adverse Events (participants affected / at risk) | 7/240
Other Adverse Events (participants affected / at risk) | 201/240
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Rimegepant 75 mg ODT (N=240)
Arteriosclerosis coronary artery (Cardiac disorders) | 1
Pneumonia (Infections and infestations) | 1
Clavicle fracture (Injury, poisoning and procedural complications) | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1
Benign breast neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Brain injury (Nervous system disorders) | 1
Varicose vein (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Rimegepant 75 mg ODT (N=240)
COVID-19 (Infections and infestations) | 100
Upper respiratory tract infection (Infections and infestations) | 28
Nasopharyngitis (Infections and infestations) | 17
Urinary tract infection (Infections and infestations) | 7
Influenza (Infections and infestations) | 6
Pharyngitis (Infections and infestations) | 6
Respiratory tract infection (Infections and infestations) | 6
Hyperuricaemia (Metabolism and nutrition disorders) | 18
Hyperlipidaemia (Metabolism and nutrition disorders) | 16
Weight increased (Investigations) | 11
Weight decreased (Investigations) | 9
Alanine aminotransferase increased (Investigations) | 7
Aspartate aminotransferase increased (Investigations) | 6
Blood creatine phosphokinase increased (Investigations) | 5
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 10
Cough (Respiratory, thoracic and mediastinal disorders) | 9
Sinus arrhythmia (Cardiac disorders) | 9
Sinus bradycardia (Cardiac disorders) | 6
Pyrexia (General disorders) | 13
Hepatic function abnormal (Hepatobiliary disorders) | 10
Anaemia (Blood and lymphatic system disorders) | 9
Toothache (Gastrointestinal disorders) | 8
Insomnia (Psychiatric disorders) | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publication until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2023-09-07): https://cdn.clinicaltrials.gov/large-docs/52/NCT05371652/Prot_000.pdf
  • Statistical Analysis Plan (2024-09-10): https://cdn.clinicaltrials.gov/large-docs/52/NCT05371652/SAP_001.pdf